CLINICAL TRIAL: NCT03312426
Title: Randomized, Open-Label Study to Assess the Effect of a Light Meal and a High-Fat Meal on the Bioavailability of a Single 100-mg Dose of BMS-986205 Commercial Tablet in Healthy Participants
Brief Title: An Investigational Study to Assess the Effect of a Light Meal and a High-Fat Meal on the Absorption of BMS-986205 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CA017-053
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: Cancer; Tumor; Healthy Participants; Healthy Subjects; Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — linrodostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986205 under fasted conditions then with high-fat meal. (Experimental): Single, 100 mg dose of BMS-986205 under fasted conditions (Day 1) followed by single, 100 mg dose of BMS-986205 with a high-fat meal (Day 15).
  Interventions: Drug: BMS-986205
- BMS-986205 with high-fat meal then under fasted conditions. (Experimental): Single, 100 mg dose of BMS-986205 with a high-fat meal (Day 1) followed by single, 100 mg dose of BMS-986205 under fasted conditions (Day 15).
  Interventions: Drug: BMS-986205
- BMS-986205 under fasted conditions then with light meal. (Experimental): Single, 100 mg dose of BMS-986205 under fasted conditions (Day 1) followed by single, 100 mg dose of BMS-986205 with a light meal (Day 15).
  Interventions: Drug: BMS-986205
- BMS-986205 with light meal then under fasted conditions. (Experimental): Single, 100 mg dose of BMS-986205 with a light meal (Day 1) followed by single, 100 mg dose of BMS-986205 under fasted conditions (Day 15).
  Interventions: Drug: BMS-986205

INTERVENTIONS:
Drug: BMS-986205 — Single dose, 100 mg administered at Day 1 and at Day 15.

SUMMARY:
The purpose of this study is to investigate the effect of a light meal and a high-fat meal on the bioavailability (absorption) of of BMS-986205 commercial tablet in healthy participants. Eligible participants will receive a single dose of BMS-986205 under fasted or fed (high-fat meal or light meal) conditions on Day 1 and Day 15. The safety, tolerability and movement of the BMS-986205 into, through and out of the body (pharmacokinetics/PK) under these conditions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent form.
* Healthy male and female participants (not of childbearing potential), determined by no clinically significant deviation from normal in medical history, physical examination, ECGs (electrocardiograms), and clinical laboratory determinations.
* Women participants must have documented proof they are not of childbearing potential.
* Males sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for duration of treatment with BMS-986205, and for a total of 110 days after the last dose of BMS-986205; and must be willing to refrain from sperm donation during this time. Azoospermic males are exempt from contraceptive requirements.
* Normal renal function at screening (Glomerula Filtration Rate ≥ 80 mL/min/1.73 m2.
* Body Mass Index (BMI) of 18.0 kg/m2 to 32.0 kg/m2 inclusive.

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding.
* Any significant acute or chronic illness.
* Active tuberculosis (TB) requiring treatment, documented latent TB within the previous 3 years, or evidence of a past TB infection without documented adequate therapy. All participants will be required to have a QuantiFERON-TB Gold test performed at screening.
* History of Glucose-6-Phosphate Dehydrogenase deficiency (G6PD) or any other congenital hemolytic anemias.
* History of cardiac arrhythmias and/or autonomic instability.
* History of pulmonary, renal or liver disease.
* History of Gilbert's Syndrome.
* Recent (within 6 months of study drug administration) history of smoking or current smokers, including use of electronic cigarettes or nicotine-containing products such as tobacco for chewing, nicotine patches, nicotine lozenges or nicotine gum.
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo or psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger may enroll.
* Major surgery within 4 weeks of study drug administration.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) following administration of single, 100 mg tablet of BMS-986205 with a high-fat meal. | Up to 21 days
  Measured by plasma concentration.
Area under the plasma concentration-time curve from time zero to 168 hours (AUC[0-168]) following administration of single, 100 mg tablet of BMS-986205 with a high-fat meal. | Up to 21 days
  Measured by plasma concentration.
Cmax following administration of single, 100 mg tablet of BMS-986205 with a light meal. | Up to 21 days
  Measured by plasma concentration.
AUC(0-168) following administration of single, 100 mg tablet of BMS-986205 with a light meal. | Up to 21 days
  Measured by plasma concentration.

SECONDARY OUTCOMES:
Number of participants with non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs) following administration of single, 100 mg tablet of BMS-986205 under fasting conditions, with a light meal or with a high-fat meal. | Day 1 up to Day 22
  Safety and tolerability of BMS-986205 measured by investigator assessment.
Results of clinical laboratory tests | Up to 22 days
  Measured by Investigator assessment
Results of vital sign measurements | Up to 22 days
  Measured by Investigator assessment
Results of electrocardiogram (ECG) | Up to 22 days
  Measured by Investigator Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Austin Clinic, Austin, Texas, United States

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx